CLINICAL TRIAL: NCT05471570
Title: The Effect of tDCS Stimulation of Right Inferior Frontal Gyrus on Language Recovery in Speakers With Aphasia
Brief Title: Effect of Anodal Transcranial Direct Current Stimulation (tDCS) Over the Right-hemisphere on Picture Naming in Chronic Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Mehdi Bakhtiar, Assistant professor, The University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: tDCSAphasia
Record Dates: First submitted 2022-07-18; First posted 2022-07-25 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Aphasia
Keywords: tDCS; Aphasia; naming
MeSH Terms: conditions — Aphasia | interventions — Transcranial Direct Current Stimulation; Language Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- anodal tDCS (Active Comparator): 20 minutes of one mA anodal High-Definition tDCS (HD-tDCS) over right IFG combined with 40 minutes of naming therapy for five consecutive days in week 1
  Interventions: Device: tDCS stimulation
- sham tDCS (Sham Comparator): 20-minutes sham HD-tDCS with 40-minutes therapy of naming therapy for five consecutive days in week 1
  Interventions: Device: tDCS stimulation

INTERVENTIONS:
Device: tDCS stimulation — The study examines the effect of excitatory stimulation of right inferior frontal gyrus (IFG) on naming abilities of people with aphasia (PWA) as compared to sham stimulation to examine the compensatory versus interference role of right hemisphere in language recovery after stroke.
  Other Names: language therapy

SUMMARY:
There are two opposing hypotheses, namely the interference and laterality-shift hypotheses, regarding the role of the right hemisphere (RH) in language recovery following a left hemisphere damage. Transcranial direct current stimulation (tDCS) has received increasing attention as a potential complement to behavioural therapy.

This preliminary study aimed to examine the effect of excitatory (anodal) stimulation of right inferior frontal gyrus (IFG) on naming abilities of chronic people with aphasia (PWA) to examine the compensatory versus interference role of RH in language recovery, and to confirm the application of tDCS does not induce adverse effects on other cognitive and language functions.

ELIGIBILITY:
Inclusion Criteria:

* People with chronic aphasia following the stroke

Exclusion Criteria:

* history of seizure or epilepsy,
* previous adverse reactions to TMS/tDCS,
* having a pace-maker or a metal implanted in the brain
* being pregnant

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Picture naming task | Immediately after the end of each treatment session and block
  One hundred and sixty pictures of concrete nouns from the Snodgrass and Vanderwart (1980) picture set (colored version) were utilised to measure the percentage of object naming accuracy. In particular, these pictures were divided into Set A (training targets) and Set B (untrained generalization targets), with eighty stimuli in each set.

SECONDARY OUTCOMES:
language task | Immediately after the end of each treatment block
  * Overall language skills are measured through the overall aphasia scores provided by the Cantonese version of Western Aphasia Battery (short-form).
  The scale is called Aphasia quotient: Minimum value = 0, maximum value = 100, with higher scores mean a better performance.
Cognitive task | Immediately after the end of each treatment block
  The cognitive skills are measured through the subtest scores provided by Oxford Cognitive Screening-Cantonese. The test uses different sub-tests including the Picture naming, Semantics, Orientation, Visual field task, Sentence reading , Calculation, Attention, Praxis, Memory, and Executive tasks. The range of values varies across the subtests. For all subtests except the executive task, the higher scores reflect better performance. For executive tasks the lower scores reflect better performance.

IPD SHARING:
Plan to Share IPD: No